CLINICAL TRIAL: NCT02128295
Title: Randomised Trial Comparing the Efficacy and Acceptability of Two Single Electric Breast Pump in Mothers Exclusively Breast Feeding Their Healthy Term Infants.
Brief Title: Trial of Two Electric Breast Pumps in Mothers of Term Infants.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Northwell Health (Other); Scientific Center of Children (Unknown); Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12NT04; UCL Ethics project ID 5645/001 (Other: UCL Ethics)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-10

CONDITIONS: Volume of Breast Milk Expressed Using Single Electric Breast Pumps.; Duration of Exclusive Breast-feeding; Duration of Any Breast-feeding
Keywords: Breast pumps, breast milk, expression, term infants
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primiparous mothers (Experimental): Mother who are primiparous
  Interventions: Device: Electric breast pump - A; Device: Electric breast pump - B
- Multiparous mothers (Experimental): Mothers who are multiparous
  Interventions: Device: Electric breast pump - A; Device: Electric breast pump - B

INTERVENTIONS:
Device: Electric breast pump - A
  Other Names: Philips Avent single electric breast pump
Device: Electric breast pump - B
  Other Names: Medela Swing single electric breast pump

SUMMARY:
This is a randomised trial of two modern single electric breast pumps allocated to mothers who are exclusively breast feeding their healthy term infants. Mothers will be recruited when their infants are around a month old, they will be randomised either to use one of two state of the art modern single electric breast pumps or to act as controls with no breast pump (but will receive a baby care voucher of similar value). If allocated to a breast pump, mothers will be asked to take part in a physiological study when their babies are 6 weeks old. In this test the mothers will be asked to express breast milk for 10 minutes on each breast. The primary hypothesis is that the total weight of milk produced in a 20 minute period and the weight of milk produced at 1 minute intervals at age 6 weeks will be greater for mothers using one of the pumps. A small sample of breast milk (~5ml) will be collected for analysis, the remaining expressed milk will returned to the mother.

Each month between the age of 3 and 6 months, all the mothers will be asked to complete online questionnaires about their breast-feeding and the use of their breast pumps (if they have one). At the end of the six months the mothers will be given a small voucher for a child-care store as a way of saying 'thank-you' for the inconvenience caused.

ELIGIBILITY:
Inclusion Criteria:

Mothers who have delivered healthy, term, singleton infants with no contra-indications for successful breast feeding.

Mothers who are exclusively breast feeding and are willing to be randomised to either use a breast pump or to continue breastfeeding without using a breast pump.

Not already using a breast pump. Can speak, read and write in English (or Chinese for Beijing centre or Russian for Moscow centre)

Exclusion Criteria:

Mothers are ineligible to join the study:

If they are mixed or formula feeding. Have an illness that may prevent them from expressing breast milk. Are not willing to be randomly assigned to the pump or the control group Already expressing milk regularly.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
The total weight of milk expressed in a set 20 minute period (10 minutes / breast) | up to 20 minutes
  The weight of milk expressed will be measured every minute for 20 minutes (10 mins/side) when the infants are around 5-6 weeks old.

SECONDARY OUTCOMES:
Exclusive and partial breast-feeding | up to 6 months
  Data will be collected at the end of each month when infants are 3 to 6 months of age to record if the infants are still being exclusively or partially breast-fed.

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Fewtrell, MD, Principal Investigator — Institute of Child Health, UCL London
Locations (1):
- Nutrition Unit, ICH-UCL, London, London, United Kingdom